CLINICAL TRIAL: NCT04647318
Title: Physiological Response to Self-compassion Versus Relaxation in a Clinical Population
Brief Title: Physiological Response to Self-compassion Versus Relaxation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Los Andes, Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UT-PSI000104
Record Dates: First submitted 2020-10-27; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Depression; Anxiety Disorders
Keywords: Compassion; Heart-rate variability; Self-criticism
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compassion focused imagery, relaxation imagery and control task (Experimental): Participants engage in three tasks (compassion focused imagery, relaxation imagery and control task), three or four times every three days.
  Interventions: Behavioral: Compassion focused imagery, relaxation imagery and control task

INTERVENTIONS:
Behavioral: Compassion focused imagery, relaxation imagery and control task — Participants will engage in three tasks (control task, relaxation imagery, and CFI) every three days on a total of 3-4 occasions. Audio-recordings of scripts will be used for both relaxation and compassion imagery. The 4-minute relaxation imagery will involve the following components (i) breathing deeply and bringing mindful awareness to the breath, (ii) relaxing the body, (iii) multisensory mental imagery of a beach or a forest, (iv) noticing feelings that arise. The 4-minute self-compassion imagery scripts will involve the following components: (i) informing participants that showing ourselves self-compassion is an effective emotional-regulation tool, (ii) breathing deeply and attending mindfully to the breath, (iii) imagining oneself embodying the four characteristics of compassion according to Gilbert5, (iv) imagine wishing oneself free of suffering using a warm voice tone and (v) noticing feelings that arise. The control task will involve reading a local city culture magazine.

SUMMARY:
Compassion-focused imagery (CFI, in which one imagines receiving or giving compassion) can be an effective emotion-regulation technique but some individuals respond as if it is a threat. However, these findings have been based on tasks involving receiving compassion from others. This study sought to examine whether CFI involving self-compassion is less threatening than relaxation and whether any threat-responses decrease with practice. This study will compare the effects of CFI, relaxation and a control task and will explore their effects on self-report symptoms and physiology. It is hypothesized that CFI involving self-compassion is less threatening than relaxation and that any threat-responses decrease with practice.

DETAILED DESCRIPTION:
Introduction

Self-criticism represents a crucial phenomenon in a variety of mental disorders1. Highly self-critical individuals show a poorly regulated threat emotional system and underdeveloped capacities for emotional regulation2,3. Self-criticism is considered a vulnerability risk factor for most psychopathological conditions. Several interventions aiming at increasing compassion as an antidote to self-criticism have been developed4. One of the most empirically validated is Compassion Focused Therapy (CFT, 5), which aims to increase acceptance and compassion for one's own suffering in order to generate a self-soothing response6.

Compassion-focused imagery (CFI) is a key technique in CFT, which involves visualizing compassion towards others, or imagining people, places or objects directing compassion towards oneself7. Single trials of CFI have shown a reduction of negative affect, an increase in self-esteem, and physiological changes associated with the attenuation of threat-focused behaviors8-10. Regular CFI practice has increased self-compassion and reduced negative affect in clinical and non-clinical populations10-13. Despite these promising findings, CFI can create threat-focused responses in some individuals; however, these findings have been based on tasks involving receiving compassion from others.

This study will explore two empirical questions:

1. How do clinical participants initially respond to self-compassionate imagery in an initial trial? The investigators hypothesize that CFI and relaxation imagery would be associated with similar levels of HRV, and that both would be associated with higher HRV than during the control task (both in terms of group means and number of people showing clinically-significant changes). It is also hypothesized that some participants would show reliable increase in positive affect and reliable decrease in negative affect during CFI, but that others would show the opposite pattern (due to inhibitors of compassion).
2. Do any threat responses reduce following repeated trials of self-compassionate imagery? It is hypothesized that the number of individuals responding negatively to CFI would decrease over time.

Methods

Participants will complete an initial screening questionnaire online that consists of reading the study information and completing informed consent, demographics questions, ODSIS14, OASIS15 and FSCRS16. Eligible participants will be invited to attend in-person sessions, in which physiological and self-report responses will be collected. Participants will be asked to avoid exercising, drinking alcohol/caffeine, smoking nicotine and eating during the two hours prior to each session, since these are possible confounds to HRV measurements. Participants will also be asked each session to confirm that they have not made any medication changes, in line with inclusion criteria. HRV will be measured by a research assistant whilst the participant engages in three 4-minute activities, always in the following order: (i) reading a local city culture magazine (control task), (ii) engaging in relaxation imagery involving walking through a forest or on a beach, and (iii) engaging in self-compassion imagery.

Participants will be randomized to complete 3 or 4 trials using a 2:1 ratio. This was decided based upon the premise that more trials are helpful for answering the research questions regarding the impact of repeated trials, but also aiming to minimize dropout for a related study which explored the effects of psychotherapy which was offered following these 3-4 trials.

Although no study to date has explored the hypotheses of this study, the investigators have set a target sample of N=25 based upon other studies exploring effects of CFI on physiology, which have samples ranging from 22 to 25 participants and found significant between-group differences in physiological measures during CFI10,17.

Data analysis

The data will be uploaded to Open Science Framework. Paired sample t-tests will be used to explore differences in RMSSD HRV during the three tasks, and to test changes in positive and negative affect from pre- to post-CFI.

To complement group-level analyses, the investigators will use reliable or clinically-significant change analyses of individuals. A reliable change index (RCI,18) will be calculated for positive and negative affect. Each participant´s change scores (calculated by subtracting pre-CFI affect from post-CFI affect for each trial) will be compared against the RCIs. The investigators will also calculate how many individuals show a clinically-significant HRV response, defined as 5ms change in RMSSD during the experimental task (CFI or relaxation) compared to the control task. THis value was based upon literature on the differences in baseline levels of HRV between healthy controls and patients with depression19,20. The number of positive and negative clinically-significant responses will be compared (i) between relaxation and compassion at trial 1 in order to compare effects of both tasks, and (ii) over 3-4 trials for both relaxation and for compassion, to evaluate whether repeated trials improved response to each task.

Attrition and data loss

Participants will be included if they complete at least one trial of the three tasks, since they can still inform the research questions focused on the initial trial data. Participants will be excluded if HRV data at trial 1 is not interpretable, as this is the primary outcome measure. Individual HRV measurements will be excluded from analysis if the participant reports any of the external threats to HRV data validity mentioned above (e.g. medication changes, high caffeine use, exercise)

ELIGIBILITY:
Inclusion Criteria:

* Being ≥18 years old
* A clinical level of depression or anxiety (defined as ≥ 8 on the ODSIS14 or OASIS15)
* High self-criticism or low self-reassurance, as measured by the FSCRS16 (≥24 on self-inadequacy, ≥ 8 on self-hatred, or ≤18 on self-reassurance). These cut-offs correspond to 0.5 SD above the mean in self-inadequacy/self-hatred, and 0.5 SD below the mean on self-reassurance, based on a validation of the FSCRS17 in Colombia28.

Exclusion Criteria (Note: these were added subsequent to seeking ethical approval but before study commencement):

* Positive screen on the Mood Disorder Questionnaire (MDQ), following the norms published by the authors
* Positive screen on the Standardised Assessment of Personality - Abbreviated Scale (SAPAS), defined as scoring 4+
* Severity of Dependence Scale (SDS): scoring 3+ for alcohol use or 5+ for other substances.
* Significant suicidal ideation. Participants were asked, "On a scale of 1 to 7, what is your intent to end your life right now?" from 1 (low) to 7 (high), and "Are you uncertain about being able to control suicidal impulses?" (Yes/No). Participants were excluded for responding ≥5 on item 1 or "yes" to item 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Difference in heart rate variability (HRV RMSSD) between three tasks: compassion, relaxation, control. | Session 1 (day 1)
  The physiological measurement system BIOPAC MP15024 will be used to collect ECG data during each task. A standard electrode configuration will be used for collecting ECG data. The ECG signal will be digitized at 2000 Hz and inspected offline using Kubios software25. Successive R waves (identified by an automatic beat detection algorithm) will be visually inspected, and any irregularities will be edited. A time domain index of HRV (RMSSD) will then be obtained for baseline, induction and each experimental condition using HRV Analysis Software26. RMSSD has been chosen because, according to the Task Force guidelines27, it reflects the integrity of vagus nerve-mediated autonomic control of the heart. Additionally, clinically-significant change can be calculated for this.
Difference in heart rate variability (HRV RMSSD) between three tasks: compassion, relaxation, control. | Session 2 (day 4)
  The physiological measurement system BIOPAC MP15024 will be used to collect ECG data during each task. A standard electrode configuration will be used for collecting ECG data. The ECG signal will be digitized at 2000 Hz and inspected offline using Kubios software25. Successive R waves (identified by an automatic beat detection algorithm) will be visually inspected, and any irregularities will be edited. A time domain index of HRV (RMSSD) will then be obtained for baseline, induction and each experimental condition using HRV Analysis Software26. RMSSD has been chosen because, according to the Task Force guidelines27, it reflects the integrity of vagus nerve-mediated autonomic control of the heart. Additionally, clinically-significant change can be calculated for this.
Difference in heart rate variability (HRV RMSSD) between three tasks: compassion, relaxation, control. | Session 3 (day 7)
  The physiological measurement system BIOPAC MP15024 will be used to collect ECG data during each task. A standard electrode configuration will be used for collecting ECG data. The ECG signal will be digitized at 2000 Hz and inspected offline using Kubios software25. Successive R waves (identified by an automatic beat detection algorithm) will be visually inspected, and any irregularities will be edited. A time domain index of HRV (RMSSD) will then be obtained for baseline, induction and each experimental condition using HRV Analysis Software26. RMSSD has been chosen because, according to the Task Force guidelines27, it reflects the integrity of vagus nerve-mediated autonomic control of the heart. Additionally, clinically-significant change can be calculated for this.
Difference in heart rate variability (HRV RMSSD) between three tasks: compassion, relaxation, control. | Session 4 (day 10)
  The physiological measurement system BIOPAC MP15024 will be used to collect ECG data during each task. A standard electrode configuration will be used for collecting ECG data. The ECG signal will be digitized at 2000 Hz and inspected offline using Kubios software25. Successive R waves (identified by an automatic beat detection algorithm) will be visually inspected, and any irregularities will be edited. A time domain index of HRV (RMSSD) will then be obtained for baseline, induction and each experimental condition using HRV Analysis Software26. RMSSD has been chosen because, according to the Task Force guidelines27, it reflects the integrity of vagus nerve-mediated autonomic control of the heart. Additionally, clinically-significant change can be calculated for this.

SECONDARY OUTCOMES:
Change in "Safe/warmth positive affect" during compassion imagery at session 1 | Session 1 (day 1), immediately pre- and immediately post-compassion-focused imagery
  Positive affect will be measured with two items from the Safe/warmth positive affect scale (safe, content) by Gilbert and colleagues23. Each item is scored from 0-4 (thus total scores will range from 0-8) with higher scores representing greater positive affect. These will be combined with the Relaxed positive affect scale (see below) into one soothing positive affect scale if acceptable internal consistency is achieved (alpha >.80), or will be analysed as two subscales if not.
  Ref 23: Gilbert, P., McEwan, K., Mitra, R., Franks, L., Richter, A. & Rockliff, H. (2008). Feeling safe and content: A specific affect regulation system? Relationship to depression, anxiety, stress, and self-criticism. The Journal of Positive Psychology, 3, 182-191.
Change in "Safe/warmth positive affect" during compassion imagery at session 2 | Session 2 (day 4), immediately pre- and immediately post-compassion-focused imagery
  See outcome 5
Change in "Safe/warmth positive affect" during compassion imagery at session 3 | Session 3 (day 7), immediately pre- and immediately post-compassion-focused imagery
  See outcome 5
Change in "Safe/warmth positive affect" during compassion imagery at session 4 | Session 4 (day 10), immediately pre- and immediately post-compassion-focused imagery
  See outcome 5
Change in "Relaxed positive affect" during compassion imagery at session 1 | Session 1 (day 1), immediately pre- and immediately post-compassion-focused imagery
  Positive affect will be measured with two items from the Relaxed positive affect scale (calm, relaxed) by Gilbert and colleagues23. Each item is scored from 0-4 (thus total scores will range from 0-8) with higher scores representing greater positive affect. These will be combined with the items from the Safe/warmth positive affect scale into one soothing positive affect scale if acceptable internal consistency is achieved (alpha >.80), or will be analysed as two subscales if not.
  Ref 23: Gilbert, P., McEwan, K., Mitra, R., Franks, L., Richter, A. & Rockliff, H. (2008). Feeling safe and content: A specific affect regulation system? Relationship to depression, anxiety, stress, and self-criticism. The Journal of Positive Psychology, 3, 182-191.
Change in "Relaxed positive affect" during compassion imagery at session 2 | Session 2 (day 4), immediately pre- and immediately post-compassion-focused imagery
  See outcome 9
Change in "Relaxed positive affect" during compassion imagery at session 3 | Session 3 (day 7), immediately pre- and immediately post-compassion-focused imagery
  See outcome 9
Change in "Relaxed positive affect" during compassion imagery at session 4 | Session 4 (day 10), immediately pre- and immediately post-compassion-focused imagery
  See outcome 9
Change in "negative threat-focused affect" during compassion imagery at session 1 | Session 1 (day 1), immediately pre- and immediately post-compassion-focused imagery
  Negative affect will be measured with four items selected by the authors of this study to tap into threat-focused emotions (anxious, distressed, vulnerable, insecure). These were selected by the authors as no appropriate validated measure was identified. Mirroring outcomes 5-12, each item will be scored from 0 (Not Characteristic of me) to 4 (Very Characteristic of me), thus total scores will range from 0-16), with higher scores representing greater negative affect.
Change in "negative threat-focused affect" during compassion imagery at session 2 | Session 2 (day 4), immediately pre- and immediately post-compassion-focused imagery
  See outcome 13
Change in "negative threat-focused affect" during compassion imagery at session 3 | Session 3 (day 7), immediately pre- and immediately post-compassion-focused imagery
  See outcome 13
Change in "negative threat-focused affect" during compassion imagery at session 4 | Session 4 (day 10), immediately pre- and immediately post-compassion-focused imagery
  See outcome 13

CONTACTS AND LOCATIONS:
Overall Officials: Iona Naismith, DClinPsy, Principal Investigator — University of the Andes
Locations (1):
- University of the Andes, Bogotá, Colombia

REFERENCES:
- [Background] Werner AM, Tibubos AN, Rohrmann S, Reiss N. The clinical trait self-criticism and its relation to psychopathology: A systematic review - Update. J Affect Disord. 2019 Mar 1;246:530-547. doi: 10.1016/j.jad.2018.12.069. Epub 2018 Dec 25. PMID 30599378
- [Background] Gilbert P, Procter S. Compassionate mind training for people with high shame and self-criticism: overview and pilot study of a group therapy approach. Clin Psychol Psychother [Internet]. 2006 Nov;13(6):353-79.
- [Background] Krieger T, Reber F, von Glutz B, Urech A, Moser CT, Schulz A, Berger T. An Internet-Based Compassion-Focused Intervention for Increased Self-Criticism: A Randomized Controlled Trial. Behav Ther. 2019 Mar;50(2):430-445. doi: 10.1016/j.beth.2018.08.003. Epub 2018 Aug 17. PMID 30824257
- [Background] Kirby JN, Tellegen CL, Steindl SR. A Meta-Analysis of Compassion-Based Interventions: Current State of Knowledge and Future Directions. Behav Ther. 2017 Nov;48(6):778-792. doi: 10.1016/j.beth.2017.06.003. Epub 2017 Jun 21. PMID 29029675
- [Background] Gilbert P. The origins and nature of compassion focused therapy. Br J Clin Psychol. 2014 Mar;53(1):6-41. doi: 10.1111/bjc.12043. PMID 24588760
- [Background] Boersma K, Håkanson A, Salomonsson E, Johansson I. Compassion Focused Therapy to Counteract Shame, Self-Criticism and Isolation. A Replicated Single Case Experimental Study for Individuals With Social Anxiety. J Contemp Psychother [Internet]. 2015 Jun 6;45(2):89-98.
- [Background] Gilbert P. Compassion focused therapy: Distinctive features. London: Routledge; 2010.
- [Background] Lincoln TM, Hohenhaus F, Hartmann M. Can Paranoid Thoughts be Reduced by Targeting Negative Emotions and Self-Esteem? An Experimental Investigation of a Brief Compassion-Focused Intervention. Cognit Ther Res [Internet]. 2013 Apr 14;37(2):390-402.
- [Background] Petrocchi N, Ottaviani C, Couyoumdjian A. Compassion at the mirror: Exposure to a mirror increases the efficacy of a self-compassion manipulation in enhancing soothing positive affect and heart rate variability. J Posit Psychol [Internet]. 2017 Nov 2;12(6):525-36.
- [Background] Rockliff H, Gilbert P, McEwan K, Lightman S, Glover D. A pilot exploration of heart rate variability and salivary cortisol responses to compassion-focused imagery. 2008.
- [Background] Gilbert P, Irons C. A pilot exploration of the use of compassionate images in a group of self-critical people. Memory. 2004 Jul;12(4):507-16. doi: 10.1080/09658210444000115. PMID 15487546
- [Background] McEwan K, Gilbert P. A pilot feasibility study exploring the practising of compassionate imagery exercises in a nonclinical population. Psychol Psychother. 2016 Jun;89(2):239-43. doi: 10.1111/papt.12078. Epub 2015 Oct 10. PMID 26454144
- [Background] Naismith I, Mwale A, Feigenbaum J. Inhibitors and facilitators of compassion-focused imagery in personality disorder. Clin Psychol Psychother. 2018 Mar;25(2):283-291. doi: 10.1002/cpp.2161. Epub 2017 Dec 18. PMID 29251381
- [Background] Bentley KH, Gallagher MW, Carl JR, Barlow DH. Development and validation of the Overall Depression Severity and Impairment Scale. Psychol Assess. 2014 Sep;26(3):815-830. doi: 10.1037/a0036216. Epub 2014 Apr 7. PMID 24708078
- [Background] Norman SB, Cissell SH, Means-Christensen AJ, Stein MB. Development and validation of an Overall Anxiety Severity And Impairment Scale (OASIS). Depress Anxiety. 2006;23(4):245-9. doi: 10.1002/da.20182. PMID 16688739
- [Background] Gilbert P, Clarke M, Hempel S, Miles JN, Irons C. Criticizing and reassuring oneself: An exploration of forms, styles and reasons in female students. Br J Clin Psychol. 2004 Mar;43(Pt 1):31-50. doi: 10.1348/014466504772812959. PMID 15005905
- [Background] Duarte J, McEwan K, Barnes C, Gilbert P, Maratos FA. Do therapeutic imagery practices affect physiological and emotional indicators of threat in high self-critics? Psychol Psychother. 2015 Sep;88(3):270-84. doi: 10.1111/papt.12043. Epub 2014 Oct 28. PMID 25347984
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127
- [Background] Hu MX, Lamers F, de Geus EJ, Penninx BW. Differential Autonomic Nervous System Reactivity in Depression and Anxiety During Stress Depending on Type of Stressor. Psychosom Med. 2016 Jun;78(5):562-72. doi: 10.1097/PSY.0000000000000313. PMID 26910796
- [Background] Moon E, Lee SH, Kim DH, Hwang B. Comparative Study of Heart Rate Variability in Patients with Schizophrenia, Bipolar Disorder, Post-traumatic Stress Disorder, or Major Depressive Disorder. Clin Psychopharmacol Neurosci. 2013 Dec;11(3):137-43. doi: 10.9758/cpn.2013.11.3.137. Epub 2013 Dec 24. PMID 24465250
- [Background] López Cavada C, Hornillos Cárdenas T, López-Romero HY. Self-criticism: measure and Treatment. Int Soc Emot Focus Ther (ISEFT), Toronto. 2017;
- [Background] Gilbert P, McEwan K, Mitra R, Franks L, Richter A, Rockliff H. Feeling safe and content: A specific affect regulation system? Relationship to depression, anxiety, stress, and self-criticism. J Posit Psychol [Internet]. 2008 Jul;3(3):182-91.
- [Background] BIOPAC Systems, Inc., Goleta, CA, United States.
- [Background] Kubios version 3.3, 2019, Biosignal Analysis and Medical Imaging Group, University of Kuopio, Finland, MATLAB.
- [Background] Niskanen JP, Tarvainen MP, Ranta-Aho PO, Karjalainen PA. Software for advanced HRV analysis. Comput Methods Programs Biomed. 2004 Oct;76(1):73-81. doi: 10.1016/j.cmpb.2004.03.004. PMID 15313543
- [Background] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210
- [Background] Naismith I, Ferro CD, Ingram G, Leal WJ. Compassion-focused imagery reduces shame and is moderated by shame, self-reassurance and multisensory imagery vividness. Res Psychother. 2019 Jan 17;22(1):329. doi: 10.4081/ripppo.2019.329. eCollection 2019 Apr 19. PMID 32913776
- [Derived] Naismith I, Otto Scheiber CS, Gonzalez Rodriguez D, Petrocchi N. Physiological response to self-compassion versus relaxation in a clinical population. PLoS One. 2023 Feb 7;18(2):e0272198. doi: 10.1371/journal.pone.0272198. eCollection 2023. PMID 36749746

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT04647318/Prot_SAP_000.pdf